CLINICAL TRIAL: NCT03235336
Title: The China Health and Nutrition Survey
Brief Title: Associations Between Tea and Sweetened Beverage Consumptions and Hyperuricemia: The China Health and Nutrition Survey
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH); China-Japan Friendship Hospital (Other); Beijing Center for Disease Control and Prevention (Other Government); University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Other Study IDs: N1706-3431
Record Dates: First submitted 2017-07-27; First posted 2017-08-01 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Nutrition Poor
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The China Health and Nutrition Survey (CHNS), an ongoing open cohort, international collaborative project between the Carolina Population Center at the University of North Carolina at Chapel Hill and the National Institute for Nutrition and Health (NINH, former National Institute of Nutrition and Food Safety) at the Chinese Center for Disease Control and Prevention (CCDC), was designed to examine the effects of the health, nutrition, and family planning policies and programs implemented by national and local governments and to see how the social and economic transformation of Chinese society is affecting the health and nutritional status of its population. The impact on nutrition and health behaviors and outcomes is gauged by changes in community organizations and programs as well as by changes in sets of household and individual economic, demographic, and social factors.

The survey was conducted by an international team of researchers whose backgrounds include nutrition, public health, economics, sociology, Chinese studies, and demography. The survey took place over a 7-day period using a multistage, random cluster process to draw a sample of about 7,200 households with over 30,000 individuals in 15 provinces and municipal cities that vary substantially in geography, economic development, public resources, and health indicators. In addition, detailed community data were collected in surveys of food markets, health facilities, family planning officials, and other social services and community leaders.

DETAILED DESCRIPTION:
Survey Design

The survey covers nine provinces that vary substantially in geography, economic development, public resources, and health indicators. A multistage, random cluster process was used to draw the samples surveyed in each of the provinces. Counties in the nine provinces were stratified by income (low, middle, and high), and a weighted sampling scheme was used to randomly select four counties in each province. In addition, the provincial capital and a lower income city were selected when feasible. In two provinces, other large cities had to be selected. Villages and townships within the counties and urban and suburban neighborhoods within the cities were selected randomly. In 1989 to 1993 there were 190 primary sampling units, and a new province and its sampling units were added in 1997. There are about 4,400 households in the overall survey, covering some 19,000 individuals. Follow-up levels are high, but families that migrate from one community to a new one are not followed. Movement within the primary sampling units and some larger urban entities is attempted.

The first round of the CHNS, including household, community, and health/family planning facility data, was collected in 1989. Six additional panels were collected in 1991, 1993, 1997, 2000, 2004, and 2006. Since the 1993 survey, all new households formed from sample households were added. Since 1997, new households in original communities were also added to replace households no longer participating in the study. Also since 1997, new communities in original provinces have been added to replace sites no longer participating. A new province was also added in 1997 when one province was unable to participate. The dropped province returned to the study in 2000.

The Chinese Ministry of Public Health has committed to continue this project as long as outside support is provided to supplement the extensive support it already provides. The research project is truly a collaborative effort, with funding with funding, expertise, and other skills shared equally by the American and Chinese institutions in significant collaborative effort.

The Household Survey

A complete household roster has been used as a reference for subsequent blocks of questions on time allocation at home (e.g., child care, elderly care, other key home activities) and economic activities. Questions on income and time allocation probe for any possible activity each person might have engaged in during the previous year, both in and out of the formal market. Information on water sources, construction, condition of the home, and ownership of consumer durables is gathered from the respondent. Additional questions probe for all possible items the household might own. Full income from market and nonmarket activities is imputed. The detailed estimation of income that is possible using these data represents a significant advance in the measurement of income in China. Inclusion of nonmonetary government subsidies such as state-subsidized housing is an especially important advance.

Health Services Section

The health services section contains detailed data on insurance coverage, medical providers, and health facilities that the household might use under selected circumstances. Questions about accessibility, time and travel costs, and perceived quality of care are asked. Information on illnesses and on all uses of the health system during the previous month is collected for children under age 7, for adults between age 20 and 45 in 1989, and from all household members in later years. Questions on immunizations, use of preventive health services, and use of family planning services are also asked.

Individual Survey

Since 2004, all questions that have related to individual activities, lifestyle, health status, marriage and birth history, body shape, and mass media exposure, etc., have been moved to two sets of individual questionnaires: for adults age 18 and older and for children and adolescents under age 18. Children age 6 and above and all adults are asked to provide their time allocation on household chores and child care, physical activities, and soft drink and sugared fruit drink consumption. Youths age 12 and older and all adults are asked their smoking status; consumption of tea, coffee, and alcohol; diet; and activity level. Adolescents age 12 and older are asked to provide their conception of their body shape. Both adolescents age 12 and older and women under age 52 married, divorced, remarried, or widowed with children age 6 to 18 in household are asked about mass-media exposure. Women under age 52 and who are married, divorced, remarried, or widowed are asked to provide their marriage, pregnancy, and birth history and inter-generational linkages to parents and parents-in-law. Adults age 55 and older are asked to provide their daily living activities and were given a memory test.

Nutrition & Physical Examination

Three days' worth of detailed household food consumption information is collected. In addition, individual dietary intake for three consecutive days is collected for every household member, irrespective of age or relationship to the household head. Adults and children receive detailed physical examinations that included weight, height, arm and head circumference, mid-arm skinfold measurements, and blood pressure (for children age 7 and older and all adults). Limited clinical nutrition and physical functioning data have been collected since 1993. Activities of daily living and related information for older adults and a new set of physical activity and inactivity data have been added for all respondents since 1997.

Community Survey

The community questionnaire (filled out for each of the primary sampling units) collects information from a knowledgeable respondent on community infrastructure (water, transport, electricity, communications, and so on), services (family planning, health facilities, retail outlets), population, prevailing wages, and related variables.

Food Market Survey

In the first two surveys, state and free market data were collected. But by 1997, none of our communities had separate state prices, so only free market stores and large stores have been visited from then onward. In all cases, prices have been collected for a representative basket of commodities.

Health and Family Planning Facility

In 1989, 1991, and 1993, separate visits were made to obtain in-depth data in each community for every identified health service and family planning provider or facility. Information was collected concerning personnel, sources of funds, services available, prices (asked separately for insured and self-pay patients), and distance to the primary sampling units served by the facility. A separate questionnaire was administered to the local family planning official about family planning policies in the community. These were discontinued in 1997, but selected questions have been of these same personnel as part of the community questionnaire since then.

ELIGIBILITY:
Inclusion Criteria:

* reported no endocrinal and rheumatological disease at baseline
* provided valid responses regarding tea consumption, soft drink consumption, and sweetened fruit drink consumption,
* provided blood samples with valid serum uric acid data

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study analyzed the participant data from the Chinese Health and Nutrition Survey (CHNS, http://www.cpc.unc.edu/projects/china), which covered nine Chinese provinces (Heilongjiang, Liaoning, Shandong, Henan, Jiangsu, Hubei, Hunan, Guizhou, and Guangxi). The CHNS used a multistage random cluster sampling method.
Sampling Method: Probability Sample
Enrollment: 5547 (Estimated)
Dates: Start 1989-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Hyperuricemia | 1997-2009
  Serum uric acid level ≥420 μmol/L in males and ≥360 μmol/L in females

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes
URL: http://www.cpc.unc.edu/projects/china

REFERENCES:
- [Result] Popkin BM, Du S, Zhai F, Zhang B. Cohort Profile: The China Health and Nutrition Survey--monitoring and understanding socio-economic and health change in China, 1989-2011. Int J Epidemiol. 2010 Dec;39(6):1435-40. doi: 10.1093/ije/dyp322. Epub 2009 Nov 3. No abstract available. PMID 19887509
- See also: Related Info — http://www.cpc.unc.edu/projects/china